CLINICAL TRIAL: NCT00625781
Title: Randomized Controlled, Multicenter Study Evaluating Treatment of Glucose Intolerance in Pregnancy
Brief Title: Treatment of Impaired Glucose Tolerance in Pregnancy
Acronym: TIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Uppsala-Örebro Regional Research Council (Other)
Responsible Party: Principal Investigator, Helena Fadl, MD, PhD, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 061018-237; TIP protocol Medscinet
Record Dates: First submitted 2008-02-01; First posted 2008-02-28 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Impaired Glucose Tolerance; Fetal Macrosomia
Keywords: Gestational diabetes mellitus; Impaired glucose Tolerance; Pregnancy; Fetal macrosomia; Treatment; Perinatal morbidity
MeSH Terms: conditions — Glucose Intolerance; Fetal Macrosomia; Diabetes, Gestational | interventions — Insulin Aspart; Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- B2 (Experimental): IGT randomized to treatment
  Interventions: Drug: Insulin aspart and Insulin human (isophane)
- B1 (No Intervention): IGT randomized to "no treatment"

INTERVENTIONS:
Drug: Insulin aspart and Insulin human (isophane) — Insulin treatment if fasting p-glucose >5.0 mmol/l or post meal value >6.5 mmol/l according to study protocol.
  Other Names: NovoRapid FlexPen, A10AB05; Insulatard FlexPen, A10AC01
  Arms: B2

SUMMARY:
The purpose of this study is to evaluate if treatment (insulin or diet) of pregnant women with impaired glucose tolerance (75-g OGTT with a fasting P-gluc <7.0 mmol/l and 2 h P-gluc >10.0 and <12.2 mmol/l) close to normoglycemia reduces children´s birth weight and neonatal morbidity. There will be a focus on treatment according to specific goals and separate follow-up regimes for the children and women post partum.

ELIGIBILITY:
Inclusion Criteria:

* Women with 75g OGTT result : fasting capillary plasma <=7.0 mmol/l and/or 2 h value >= 12.2 mmol/l

Exclusion Criteria:

* Multiple pregnancy
* Pregestational Diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-02; Primary Completion 2012-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Perinatal morbidity and intrauterine growth | 1 year post partum

SECONDARY OUTCOMES:
Children´s future health | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Hanson, Consultant, Study Chair — Uppsala Academic Hospital , Sweden; Ingrid Östlund, MD, Principal Investigator — Region Örebro County
Locations (1):
- University Hospital Örebro, Örebro, Sweden